CLINICAL TRIAL: NCT06562634
Title: Effectiveness of Ultrasound-Guided Erector Spinae Plane Block for Postoperative Pain Control in Open Knee Surgeries
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Sameh Darwish, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ESPB in knee surgeries
Record Dates: First submitted 2024-08-14; First posted 2024-08-20 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Erector Spinae Plane Block (Experimental): The patient will be placed in a prone position. A convex-array ultrasound probe will be placed in a transverse orientation at L4 level to identify the tip of the L4 transverse process .The tip of the transverse process is centered on the ultrasound screen and the probe is then rotated into a longitudinal orientation 2-3 cm lateral to vertebral column, in which the following layers will be visible superficial to the acoustic shadows of the transverse processes: skin, subcutaneous tissue, erector spinae muscle and psoas muscle. The lumbar skin region will be sterilized, local anesthetic infiltration of the superficial tissues, an echogenic 22-G block needle is inserted in-plane to the ultrasound beam in a cranial-to-caudal direction until contact was made with the L4 transverse process. A total of 20ml bupivicaine 0.25%, and 20 ml xylocaine 1% will be injected into the ESP on the affected side.
  Interventions: Procedure: erector spinea plane block
- Morphine (Experimental): intravenous morphine will be given in a dose of 0.1-0.2mg/kg to maintain intraoperative analgesia.
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Procedure: erector spinea plane block — an echogenic 22-G block needle is inserted in-plane to the ultrasound beam in a cranial-to-caudal direction until contact was made with the L4 transverse process. Correct location of the needle tip in the fascial plane deep to erector spinae muscle is confirmed by injecting 0.5-1 ml saline and seeing the fluid lifting the erector spinae muscle off the transverse process while not distending the muscle. A total of 20ml bupivicaine 0.25%, and 20 ml xylocaine 1% will be injected into the ESP on the affected side.
  Arms: Ultrasound-Guided Erector Spinae Plane Block
Drug: Morphine Sulfate — intravenous morphine will be given in a dose of 0.1-0.2mg/kg to maintain intraoperative analgesia.
  Arms: Morphine

SUMMARY:
To estimate the efficacy of the ultrasound guided ESP block for postoperative pain control in open knee surgeries under general anesthesia.

DETAILED DESCRIPTION:
Postoperative pain is a major concern after knee surgeries. It is severe in 60% of patients and moderate in 30%. When inadequately treated, it intensifies reflex responses, which leads to cause serious complications, such as cardiovascular, pulmonary or urinary problems, thromboembolism, increased oxygen consumption, hyperdynamic circulation and hinders early physical therapy. Generally it has been assumed that adequate postoperative pain relief may reduce these complications, and improve general postoperative outcome.

In the last decade Improvements in pain management techniques have had a major impact on the practice of knee surgeries. Although there are a number of treatment options for postoperative pain, a gold standard has not been established. Patient-controlled analgesia (PCA), epi¬dural analgesia and lumbar plexus and/or sciatic blocks are the commonly used routes for pain relief after joint surgery .Each of those options has advantages and disadvantages. PCA has fewer technical problems, uniform and sustained analgesia with autonomy, however it might lead to respiratory depression, nausea and vomiting. Epidural analgesia is an efficient route for postoperative analgesia ; however it is associated with technical failures, hypotension, urinary retention, and ileus, motor block that limits ambulation, unrecognized compartment syndromes, and spinal hematoma secondary to anticoagulation.

The ultrasound-guided erector spinae plane (ESP) block is a recently described regional anesthetic technique for providing thoracic analgesia when performed at the level of T5 transverse process. Local anesthetic is injected into the fascial plane deep to the erector spinae muscle, and spreads craniocaudally over several levels can lead to effective analgesia and sensory block from T2 to T9. Local anesthetic also penetrates anteriorly through the intertransverse connective tissue and enters the thoracic paravertebral space where it can potentially block not only the ventral and dorsal rami of spinal nerves but also the rami communicantes that transmit sympathetic fibers.

ESP advantages include its simplicity, easy identifiable ultrasonographic landmarks and an endpoint for injection and low risk for serious complications as injection is into tissue plane that is distant from pleura, major blood vessels and discrete nerves.

There is clinical report of two cases shows the ESP block may be a safe, simple and effective technique for analgesia following surgery around the knee.

However, confirmation of the efficacy of ESP block in knee surgeries needs more investigation.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged from 18 to 60 years old.

  * Genders eligible for study: both sexes.
  * ASA I-II.
  * Undergo knee surgery.
  * BMI from 18 to 35 kg/m2.

Exclusion Criteria:

* • Patient refusal.

  * Patients with difficulty in evaluating their level of pain.
  * Contraindications to regional anesthesia (Bleeding disorders e.g. INR>1.5, PC<70%, platelet count<100 × 109, Use of any anti-coagulants, local infection, etc.).
  * Known allergy to local anesthetics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption during the 1st 24 h postoperative. | 24 hour postoperative
  Total morphine consumption during the 1st 24 h postoperative.

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperative
Time to first postoperative analgesic request | 24hour postoperative
Visual analogue score (0-10) | 24hour postoperative
  0: no pain 10:worst pain
Hemodynamics :heart rate (bpm) | baseline ,Intraoperative every 15 min, postoperative for 24 hr
Block failure rate. | Intraoperative &24 hour postoperative
Incidence of complications. (Nerve injury, Hematoma formation, LA toxicity, Intravascular injection | 24hour postoperative
Hemodynamics :arterial blood pressure (systolic, diastolic and mean blood pressure) in mmhg | baseline, intraoperative every 15 min, postoperative for 24 hr

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo, Egypt

REFERENCES:
- [Result] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Result] Kehlet H. Postoperative pain relief--what is the issue? Br J Anaesth. 1994 Apr;72(4):375-8. doi: 10.1093/bja/72.4.375. No abstract available. PMID 8155433
- [Result] Maheshwari AV, Blum YC, Shekhar L, Ranawat AS, Ranawat CS. Multimodal pain management after total hip and knee arthroplasty at the Ranawat Orthopaedic Center. Clin Orthop Relat Res. 2009 Jun;467(6):1418-23. doi: 10.1007/s11999-009-0728-7. Epub 2009 Feb 13. PMID 19214642
- [Result] Sinatra RS, Torres J, Bustos AM. Pain management after major orthopaedic surgery: current strategies and new concepts. J Am Acad Orthop Surg. 2002 Mar-Apr;10(2):117-29. doi: 10.5435/00124635-200203000-00007. PMID 11929206
- [Result] Chelly JE, Greger J, Gebhard R, Coupe K, Clyburn TA, Buckle R, Criswell A. Continuous femoral blocks improve recovery and outcome of patients undergoing total knee arthroplasty. J Arthroplasty. 2001 Jun;16(4):436-45. doi: 10.1054/arth.2001.23622. PMID 11402405
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Result] Ayub A, Talawar P, Gupta SK, Kumar R, Alam A. Erector spinae plane block: A safe, simple and effective alternative for knee surgery. Anaesth Intensive Care. 2019 Sep;47(5):469-471. doi: 10.1177/0310057X19877655. Epub 2019 Nov 4. No abstract available. PMID 31684742
- [Result] Karmakar MK, Ho AM, Li X, Kwok WH, Tsang K, Ngan Kee WD. Ultrasound-guided lumbar plexus block through the acoustic window of the lumbar ultrasound trident. Br J Anaesth. 2008 Apr;100(4):533-7. doi: 10.1093/bja/aen026. PMID 18344573
- [Result] Weller R, Rosenblum M, Conard P, Gross JB. Comparison of epidural and patient-controlled intravenous morphine following joint replacement surgery. Can J Anaesth. 1991 Jul;38(5):582-6. doi: 10.1007/BF03008188. PMID 1934205